CLINICAL TRIAL: NCT01586598
Title: Sensory Retraining Exercise Facilitates Sensory Recovery After Bilateral Sagittal Split Osteotomy - a Randomized Controlled Trial
Brief Title: Sensory Retraining Facilitates Sensory Recovery After Mandibular Nerve Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CGMH-IRB-100-2302A3
Record Dates: First submitted 2012-02-15; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Injury of Trigeminal Nerve; Surgery; Mandibular Prognathism
Keywords: Mandibular Nerve; Orthognathic Surgery; Sagittal Split Osteotomy; Sensory Retraining
MeSH Terms: conditions — Trigeminal Nerve Injuries; Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): No intervention will be given to this control group. Spontaneous recovery of mandibular nerve will be assessed for sensory function.
- sensory retraining group (Experimental): Sensory retraining protocol will be applied this group. Any facilitation of sensory function in mandibular nerve will be assessed.
  Interventions: Behavioral: sensory retraining protocol

INTERVENTIONS:
Behavioral: sensory retraining protocol — 1. within one month after the surgery: facial massage and physical stimulation over lower face and lip, four times (20 minutes each time) a day
  2. one to three months after the surgery: brush and physical stimulation over lower face and lip, four times (20 minutes each time) a day
  3. three to six months after the surgery: brush, pin and physical stimulation over lower face and lip, four times (20 minutes each time) a day
  Other Names: sensory retraining
  Arms: sensory retraining group

SUMMARY:
The purpose of this study is to determine whether sensory retraining exercise could improve lip numbness caused by bilateral sagittal split of mandible.

DETAILED DESCRIPTION:
The study is a prospective randomized controlled trial. The patients receiving bilateral sagittal split osteotomy and having lip numbness or paraesthesia will be included in this study. 80 patients will be included and randomized into two groups and there are 40 patients in each group. The control group is to maintain follow up in clinic and do not receive any sensory retraining exercise. The experimental group is requested to perform sensory retraining at home by themselves.

ELIGIBILITY:
Inclusion Criteria:

1. Taiwanese adult (18-40 y/o)
2. Developmental dentofacial disharmony (Class III)
3. Patients received orthognathic surgery (BSSO alone or with maxillary procedure)

Exclusion Criteria:

1. Medical condition associated with systemic neuropathy
2. Unwilling to sign informed consent
3. Congenital anomaly or acute trauma affecting the face
4. Previous facial surgery
5. Positive pain sensation at first week of post-surgery
6. Altered sensation before OGS as numbness or unusual feeling
7. Cleft lip and palate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
sensory function test | one year after surgery
  The sensory function evaluation include objective and subjective examinations as the followings:
  1. Questionnaire
  2. Visual analogue scale (VAS)
  3. Two-point discrimination (2PD)
  4. Pain detection threshold (PD) tests
  5. Touch sensory threshold

CONTACTS AND LOCATIONS:
Overall Officials: Chiung Shing Huang, PhD, DDS, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan, Taiwan